CLINICAL TRIAL: NCT01273415
Title: Usefulness of Ki67 Proliferative Index to Predict Recurrence and Benefit From Adjuvant Chemotherapy in Hormone Receptor (HR)-Positive Breast Cancer
Brief Title: Usefulness of Ki67 Index in Hormone Receptor-positive Breast Cancer
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Young-Hyuck Im, professor, Samsung Medical Center
Other Study IDs: 2010-12-049
Record Dates: First submitted 2011-01-06; First posted 2011-01-10 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
Keywords: hormone receptor-positive breast cancer; nomogram; Ki67; Effects of Chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hormone receptor-positive breast cancer: postoperative hormone receptor-positive breast cancer

SUMMARY:
Gene expression studies have identified at least four molecularly distinct subtypes of breast cancer including two biologically distinct ER-positive subtypes of breast cancer: luminal A and luminal B (with luminal B tumors having poorer outcomes than luminal A tumors). Although some luminal B tumors can be identified by their expression of HER2, the major biological distinction between luminal A and B is the proliferation signatures, including genes such as CCNB1, MKI67, and MYBL2, which have higher expression in luminal B tumors than in luminal A tumors. The high cost of gene expression profiling has limited its incorporation into general clinical practice. To date, there is no available IHC-based surrogate assay that can distinguish between luminal A and luminal B tumors. We hypothesized that the IHC determination of the Ki67 index as well as ER, PgR, and HER2 status is able to distinguish the luminal B subtype of breast cancers from the luminal A subgroup.

DETAILED DESCRIPTION:
Gene expression studies have identified five molecularly distinct subtypes of breast cancer that have prognostic value across multiple treatment settings including tow biologically distinct estrogen receptor (ER)-positive subtypes of breast cancer: luminal A and luminal B.The expression of ER-associated genes characterizes the luminal breast cancers, with luminal B tumors having poorer outcomes than luminal tumors. Although some luminal B tumors can be identified by their expression of HER2, the major biological distinction between luminal A and B is the proliferation signature, including genes such as CCNB1, MKI67, and MYBL2, which have higher expression in luminal B tumors than in luminal A tumors.Therefore, a distinction between luminal A and B tumor that is based on proliferation status among ER-positive luminal patients may be important to breast cancer biology and prognosis.

The high cost of gene expression profiling has limited its incorporation into most randomized clinical trials, and thus, DNA microarray-defined proliferation status is not used to provide prognostic information in general practice. Although the Ki67 gene may have prognostic value, evaluations of this marker in the adjuvant setting raise conflicts, and in the absence of a standardized test for Ki67, it is difficult to draw firm conclusions from trials.As a result, Ki67 cannot be used to assign patients to specific treatments or risk groups.

Yet despite great uncertainty, the panel of experts at the St. Gallen Consensus in 2009 proposed to (1) classify tumors as low, intermediate, or high in proliferative potential corresponding to Ki67 labelling index values of less than or equal to 15%, 16-30%, and more than 30%, respectively, and (2) use the Ki67 labeling index as a criterion for selecting to add chemotherapy to endocrine therapy in HR-positive BCs. Since proliferation is uniformly higher in basal-like and HER2 cancers but is variable within ER-positive cancer, the greatest practical prognostic value of proliferative index seems to be within ER-positive disease. Decisions regarding the use of adjuvant therapy in early operable breast cancer depend on an array of factors that predict prognosis and therapeutic efficacy. Multigene signatures related to cell proliferation show consistent accuracy in the clinical characterization of hormone receptor (HR)-positive BC, hence interest in biologic factors that predict the adjuvant response continues to increase.

Based on this consensus, we hypothesized that in a large patient population with a long follow-up, we could determine a cut-off value for the Ki67 labeling index that is sufficiently sensitive and specific to identify the patients with HR-positive luminal BC who will not require the addition of cytotoxic chemotherapy to endocrine treatment. In addition, a comparison of the objective significance level for Ki67 with values for other confirmed biomarkers (e.g., HER2, estrogen receptor, and histologic differentiation) may clarify the value of Ki67 as a biomarker in HR-positive luminal BCs.

ELIGIBILITY:
Inclusion Criteria:

* hormone receptor-positive breast cancer patient who received curative surgery from 2004 to 2007 at Samsung Medical Center

Exclusion Criteria:

* the patients who received neoadjuvant chemotherapy the patients whose biopsy showed DCIS the patients who were not available immunohistochemical findings the patients who were not available medical record

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: postoperative hormone receptor-positive breast cancer patients from 2004 to 2007 at Samsung Medical Center
Sampling Method: Probability Sample
Enrollment: 1070 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
to validate Ki67 index to predict recurrence | from the date of diagnosis to the date of relapse

SECONDARY OUTCOMES:
to investigate cut-off value of Ki67 index | from the date of diagnosis to the date of relapse

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hyuck Im, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Park YH, Im SA, Cho EY, Ahn JH, Woo SY, Kim S, Keam B, Lee JE, Han W, Nam SJ, Park IA, Noh DY, Yang JH, Ahn JS, Im YH. Validation and comparison of CS-IHC4 scores with a nomogram to predict recurrence in hormone receptor-positive breast cancers. Oncology. 2014;86(5-6):279-88. doi: 10.1159/000362281. Epub 2014 Jun 4. PMID 24903080